CLINICAL TRIAL: NCT06333964
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of AST-001 Followed by an Open-Label Extension Treatment Period in Children With Autism Spectrum Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of AST-001 in ASD Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astrogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AST-001P_P301_ASD
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Main study(0~12 weeks) Experimental: AST-001 Comparator: Placebo of AST-001
  Extension study(12~24 weeks) Experimental: AST-001 Comparator: AST-001
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AST-001 (Experimental)
  Interventions: Drug: AST-001
- Placebo of AST-001 (Placebo Comparator)
  Interventions: Drug: Placebo of AST-001

INTERVENTIONS:
Drug: AST-001 — AST-001, PO bid for 24weeks (dosage according to weight range)
  Arms: AST-001
Drug: Placebo of AST-001 — Placebo of AST-001, PO bid for 12 weeks + AST-001, PO bid for 12 weeks (dosage according to weight range)
  Arms: Placebo of AST-001

SUMMARY:
1. Study purpose: To demonstrate the superiority of AST-001 compared to placebo in improving core symptoms of autism spectrum disorder (ASD) in children with ASD.
2. Background: ASD is a neurodevelopmental disorder characterized by deficits in social communication and social interaction as well as restricted, repetitive patterns of behavior, interests, or activities. There are no approved medicines to treat the core symptom of ASD. Although these drugs and other psychotropic medications are associated with side effects, the use of psychotropic drugs to treat associated psychiatric comorbidities is common. AST-001 is developed to treat the core symptom of ASD.
3. Design: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 clinical trial followed by an Open-Label Extension Treatment Period

ELIGIBILITY:
Inclusion Criteria:

* Those who meet the criteria of diagnostic and statistical manual of mental disorder (DSM)-5 during screening
* During screening period, individuals who are diagnosed with ASD through ADI-R assessment
* Subject with a CGI-S score of 4 or higher as a result of Clinical Global Impression(CGI) evaluation during baseline visit(visit 2)
* Subject or/and legally authorized representative voluntarily agreed to participate in this clinical trial and provided their informed consent by signing the written consent form
* In case of subjects who were receiving non-pharmacological therapy at the time of screening, the non-pharmacological therapy lasted at least 3 months prior to participation in screening and is expected to be sustainable during this clinical trial
* Subject whose legally authorized representative is able to participate in the provision of reliable information about the subject's condition, execute all scheduled site visits, oversee IP administration, fully understand and speak Korean, and conduct survey evaluation regarding the subject

Exclusion Criteria:

* At the time of screening, subject has the medical history, concomitant condition, or surgical history
* During the screening period, uncontrolled medical conditions,
* During the screening period, display of severe self-harm or injury to others that requires medical treatment, determined by investigator
* At the time of screening, weight over 60kg
* Inappropriate to participate in the trial determined by investigator

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
K-VABS-II (Korean-Vineland Adaptive Behavior Scale-II) | Baseline, 12week, 24week

SECONDARY OUTCOMES:
CGI (Clinical Global Impression) | Baseline, 4week, 8week, 12week, 18week, 24week
SRS-2 (Social Responsiveness Scale-2) | Baseline, 4week, 12week, 24week
K-PSI-4-SF (Korean-Parenting Stress Index-4th Edition Short Form) | Baseline, 12week, 24week

CONTACTS AND LOCATIONS:
Overall Officials: Yoo-Sook Joung, MD, Ph.D, Principal Investigator — Samsung Medical Center
Locations (11):
- South Korea (11):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Hallym University Medical Center, Anyang-si, Gyeonggi-do
  - Samsung Changwon Medical Center, Changwon, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Koera University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No